CLINICAL TRIAL: NCT06186154
Title: Vitamin B12 and Folinic Acid Supplementation in Mitochondrial DNA Deletion Syndromes
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Andre Mattman, Medical Biochemist; Clinical Professor, University of British Columbia
Allocation: Not Applicable | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: H23-02541
Record Dates: First submitted 2023-12-01; First posted 2023-12-29 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Mitochondrial DNA Deletion; Macrocytosis
Keywords: Folinic Acid; Vitamin B12; Mitochondrial DNA Deletion; Macrocytosis
MeSH Terms: interventions — Leucovorin

STUDY DESIGN:
Intervention Model Description: Pilot single group study where each study subject acts as their own control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: Folinic acid (oral); Cyanocobalamin sublingual — * Vitamin B12 (also known as Cyanocobalamin) daily sublingual supplementation of 1000 mcg/day and folinic acid orally 1mg/day
  * Laboratory: Complete blood count, electrolytes, reticulocytes, creatinine, urea, alkaline phosphatase (ALP), alanine transaminase, ferritin, total homocysteine, lactate and hemoglobin A1c. Routine blood will be collected as regular standard of care with each visit. MMA will also be assessed. Peripheral serum values (CBC, B12) will serve as a representation of central micronutrient availability
  * Clinical Evaluation: the Newcastle mitochondrial disease adult scale (NMDAS)

SUMMARY:
The purpose of this single center study is to evaluate whether there is a concordant improvement in macrocytosis in patient with mtDNA deletions with established macrocytosis following a trial of Vitamin B12 and Folinic acid supplementation.

This study aims to assess if macrocytosis in patients with mtDNA deletion syndromes improve following empiric supplementation with vitamin B12 and folic acid. Complete blood counts (CBC) will be followed during this study (at initiation, 3 months, and 6 months) to assess for response in MCV to supplementation. The potential involvement of the region affected by the mtDNA deletion in mitochondrial folate-mediated transport and metabolism [5,6] may serve as the possible link between the deletion and observed macrocytosis.

Neurologic/cognitive outcomes will also be followed at the above time intervals to assess if 3-6 months of Vitamin B12/folinic supplementation is an adequate vs insufficient time to observe a change in the Newcastle Mitochondrion Disease Adult Scale (NMDAS). The value of this study is that it may produce pilot data to support empiric supplementation of B12 and folate for patients with macrocytosis and mtDNA deletion syndromes.

Disease Large single mtDNA (mitochondrial DNA) deletion syndrome is a rare inborn error of metabolism, and chronic progressive external ophthalmoplegia (CPEO) is the most common phenotype in adults with this form of mitochondrial deletino syndrome. Upon recent review of cases from our Adult Metabolic Diseases Clinic (AMDC), several patients with mtDNA deletion syndromes (as opposed to mtDNA missense mutations identified over the same 2016-2022-year period) were found to have unexplained macrocytosis and this is the relevant study population for this assessment.

Intervention Participants will be followed as a single group for this pilot study. The study will include two phases; 6 months without micronutrient supplementation, followed by 6 months of folinic acid and B12 supplementation. Subjects will have bloodwork to establish baseline complete blood count (macrocytosis with/without anemia) as well as at 3 and 6 months without supplementation to establish a trend in the hematologic parameters above. Participants will also complete a baseline Newcastle Mitochondrion Disease Adult Scale (NMDAS) prior to supplementation, as well as at 3 and 6 months of starting supplementation. This next phase of folinic acid and B12 supplementation will continue for 6 months with biomarker monitoring again at 9 and 12 months, and the same biochemical investigations will take place to assess if there was a true association between peripheral serum macrocytosis and nutrient supplementation during the time periods.

Phase

1

DETAILED DESCRIPTION:
Study Design:

* Study type: Pilot single group study
* Actual Enrollment: 25 participants
* Allocation: N/A
* Intervention Model: Single Group Assignment
* Intervention Model Description:

  * Vitamin B12 (also known as Cyanocobalamin) daily sublingual supplementation of 1000 mcg/day and folinic acid orally 1mg/day
  * Laboratory: Complete blood count, electrolytes, reticulocytes, creatinine, urea, alkaline phosphatase (ALP), alanine transaminase, ferritin, total homocysteine, lactate and hemoglobin A1c. Routine blood will be collected as regular standard of care with each visit. MMA will also be assessed. Peripheral serum values (CBC, B12) will serve as a representation of central micronutrient availability
  * Clinical Evaluation: the Newcastle mitochondrial disease adult scale (NMDAS)
* Masking: None (Open Label)
* Primary Purpose:

  * Assess for the proportion of subjects whose macrocytosis corrects (MCV, measured in fL, returns to the normal range of the testing laboratory) with Vitamin B12 and folinic acid supplementation in patient population with mtDNA deletion syndrome
  * Follow the Newcastle mitochondrial disease adult scale (NMDAS) with Vitamin B12 and folinic acid supplementation in patient population with mtDNA deletion syndromes for any clinical evidence of change.

The NMDAS has a maximum score of 140 (sections I, II (excluding question 8), and III). A higher score indicates more severe disease.

ELIGIBILITY:
Inclusion Criteria:

* Ages eligible for study: 19 years and older (Adult, Older Adult)
* All subjects reviewed previously at the Adult Metabolic Diseases Clinic with clinical features characteristic of major mtDNA deletion cases with biochemical macrocytosis
* Continue prior administration of other therapies pertaining to their necessary medical care
* Subjects must be clinically stable for more than one month after any stroke-like episodes
* Written, informed consent to participate in the study

Exclusion Criteria:

* Subjects with mitochondrial disease with a genetic etiology other than a major mtDNA deletion
* Palliative care patients
* Patients with a progressive neurologic disorder clinically attributable to a cause other than mitochondrial disease (e.g., ischemic stroke due to embolism from atrial fibrillation, atherosclerosis, malignant hypertension,)
* Subjects who decline blood test and/or the follow-up schedule
* Inability or refusal to give informed consent
* Coexisting participation with other investigational drug study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Macrocytosis | 1 year
  • Proportion of patients who normalize their MCV (measured in fL) such that the MCV Is within the normal range of the testing laboratory after 6 months of vitamin therapy

SECONDARY OUTCOMES:
Newcastle mitochondrial disease adult scale (NMDAS) | 1 year
  NMDAS scores (sections I-III with the exception of question 8 in section II) at scheduled intervals to assess for any clinically-evident change following supplementation introduction. Total score 140. Higher score indicates more severe disease

IPD SHARING:
Plan to Share IPD: No